CLINICAL TRIAL: NCT05825586
Title: An Interventional, Non-comparative, Single-center Post Marketing Clinical Follow-up (PMCF) Study to Evaluate Performance and Safety of "Distilled Waters-based Eyedrops" Used to Relieve Dry Eye Symptoms
Brief Title: PMCF Study to Evaluate Performance and Safety of "Distilled Waters-based Eyedrops" Used to Relieve Dry Eye Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C.O.C. Farmaceutici S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COC-R2-DW
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Dry Eye; Dry Eye Disease; Kerato Conjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eyedrops treatment arm (Experimental)
  Interventions: Device: Distilled waters based eye drops

INTERVENTIONS:
Device: Distilled waters based eye drops — Distilled Waters (DW)-based eyedrops

SUMMARY:
Dry eye disease (DED), also called keratoconjunctivitis sicca, is a common ocular condition characterized by a loss of homeostasis of the tear film and inflammation of the ocular surface. The typical symptoms of DED include irritation, discomfort, blurred or fluctuating vision.

Over the counter (OTC) artificial tears are typically the first line of dry eye treatment; they are meant to supplement the tears that cover the eye's surface. OTC products mimic the different layers of the tear film in order to maintain ocular hydration.

Distilled waters of natural herbs such as Green Tea, Calendula, Chamomile, Hamamelis and Euphrasia are known for their soothing and refreshing properties. Thanks to the combined action of these natural elements, distilled waters-based eyedrops are particularly indicated to relieve eye dryness, irritation and redness of the eyes' mucosa caused by atmospheric agents, environmental factors, and/or use of contact lenses.

"Distilled waters-based eyedrops" medical devices are ophthalmic solutions containing distilled waters able to relieve eye discomfort thanks to their soothing and refreshing action.

For these reasons, an interventional, non-comparative, single-center Post Marketing Clinical Follow-up (PMCF) study was planned to evaluate the performance and safety of "Distilled waters-based eyedrops" used as intended to relieve dry eye symptoms.

The objectives of the PMCF study are confirmation of the performance, collection of additional safety data regarding expected adverse events and detection of potential unexpected adverse events associated with use of "Distilled waters-based eyedrops" according to the IFU.

Each subject, after signing the Informed Consent Form, will enter the screening and baseline phase (the 2 visits will coincide) during which baseline procedures will be completed.

At baseline visit (V0), one of the "Distilled waters-based eyedrops" products will be administered to the enrolled subject.

The patient will perform 2 on site visits (V0 and V2/EOS). To monitor the safety, 1 phone contact is planned (V1) to check for potential adverse events and concomitant medications intake.

The first administration and the intervals at which the treatment should be repeated, to be done as per Investigator judgment and according to the IFU, depend on various factors regarding the physiology of the patients (e.g. type of eye-tear film, anatomy, age), their lifestyle (e.g. use of computer, wearing of contact lenses).

ELIGIBILITY:
Inclusion Criteria:

* Patient informed consent form (ICF) signed;
* Male and Female aged ≥ 18 years at the time of the signature of ICF;
* Patients with ophthalmic discomfort due to atmospheric agents and/or environmental factors, contact lenses wearing or dry eye symptoms;
* Willing not to use other eye drops during the entire treatment period.

Exclusion Criteria:

* Other - different - eyes clinical conditions (e.g. glaucoma);
* Suspected alcohol or drug abuse;
* Known hypersensitivity or allergy to IP components;
* Other clinically significant and uncontrolled pathologies that may interfere with study results (e.g. rheumatic diseases; diabetes);
* Participation in another investigational study;
* Inability to follow all study procedures, including attending all site visits, tests and examinations;
* Mental incapacity that precludes adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Change in Schirmer Test I: to evaluate the performance of "DW-based eyedrops" used as intended to relieve eye mucosa' irritation and redness due to atmospheric agents, environmental factors, and/or use of contact lenses, through Schirmer I test | From baseline (V0 = Day 0) at 1 month (EOS/V2 = Day 30)

SECONDARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI): to evaluate the performance of the "DW-based eyedrops" used as intended to ensure relief from eye discomfort sensation (e.g. eye strain, dryness, itching, and burning), through OSDI | From Baseline (V0 = Day 0) at 1 month (EOS/V2 = Day 30)
To evaluate the safety and tolerability of the "Distilled waters-based eyedrops" through Visual Analogue Scale (VAS) - evaluation of symptoms related to dry eye disease (burning, fatigue, discomfort, redness). | End of study visit (EOS/V2 = Day 30)
  Visual Analogue Scale:
  Minimum value = 0; Maximum value = 10; Higher scores mean a better outcome.
To evaluate the patient satisfaction of the "DW-based eyedrops" through a 5-points Likert Scale | End of study visit (EOS/V2 = Day 30)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Policlinico Mater Domini - Università Magna Grecia di Catanzaro, Catanzaro, CZ, Italy